CLINICAL TRIAL: NCT05938673
Title: Effects of Repetitive Trans Spinal Magnetic Stimulation Associated With Treadmill Gait Training on Gait Disorders in Patients With Parkinson's Disease
Brief Title: Effects of rTSMS Associated With Treadmill Training in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 57119022.4.1001.0068
Record Dates: First submitted 2023-06-02; First posted 2023-07-10 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic
Keywords: Non-invasive brain stimulation; Parkinson's disease; Spinal cord stimulation; gait
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel, phase III clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and examiners will be blinded to stimulation status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham repetitive transpinal magnetic stimulation (Sham Comparator): In the Sham group a coil will be positioned in the T2-T3 thoracic region disconnected to the stimulation device and the active coil will be positioned about 15 cm behind the patient, away from his field of vision, to provide sound stimulus.
  Interventions: Other: Sham stimulation
- Active repetitive transpinal magnetic stimulation (Active Comparator): In the Active group, the patient will receive intermittent theta burst stimulation (iTBS) in the T2-T3 region while seated using a circular magnetic coil positioned at 90º, handle facing to the right, connected to a magnetic stimulator.
  Interventions: Other: Active stimulation- intermittent theta-burst (iTBS) stimulation

INTERVENTIONS:
Other: Active stimulation- intermittent theta-burst (iTBS) stimulation — During active stimulation, patients will receive intermittent theta-burst (iTBS) stimulation in T2-T3 toracic region while seated using a circular magnetic coil positioned at 90º, handle facing to the right, connected to a magnetic stimulator.Each participant will receive a total of 1,200 rTsMS pulses at 120% of resting motor threshold, determined by abdominal muscle contractions. In 3 minutes and 58 seconds, 20 trains with 20 bursts and each burst with 3 pulses at 50 Hz repeated at 5Hz with an intertrain interval of 8 seconds will be applied.Immediately after, participants will proceed with 30 minutes of treadmill training, starting at 80% of the comfortable walking speed. Progressive speed increments of 0.2 km/h will be performed every 5 minutes as tolerated. The intensity of the exercise will be adjusted to the patient's tolerance and maintained between light to moderate intensity.
  Arms: Active repetitive transpinal magnetic stimulation
Other: Sham stimulation — During sham stimulation, a circular magnetic coil will be positioned in the T2-T3 toracic region disconnected to the stimulation device and the active coil will be positioned about 15 cm behind the patient, away from his field of vision, to provide sound stimulus. To create a sensation of muscle contraction and impression of active stimulation, the group will be submitted to the sensory effect of transcutaneous electrical neurostimulation (TENS) for 5 minutes, with surface electrodes placed in parallel at the T2-T3, with the parameters (80Hz,150ms, 60 mA).Immediately after, participants will proceed with 30 minutes of treadmill training, starting at 80% of the comfortable walking speed. Progressive speed increments of 0.2 km/h will be performed every 5 minutes as tolerated. The intensity of the exercise will be adjusted to the patient's tolerance and maintained between light to moderate intensity.
  Arms: Sham repetitive transpinal magnetic stimulation

SUMMARY:
Gait changes appear and become the main cause of disability, loss of independence, falls, fractures and reduced quality of life for patients with Parkinson Disease. Optimal gait management is complex and challenging. Some characteristics, such as gait variability, postural instability, and postural changes, continue to worsen over time despite optimal dopaminergic treatment, suggesting that additional interventions are needed. Given the physiology of gait and postural control in humans, spinal cord stimulation is a potential target for neuromodulatory approaches to gait and postural disorders. Repetitive transspinal magnetic stimulation ( rTSMS) has attracted a lot of attention, due to the possibility of modulating motor and sensory networks in a non-invasive way, activating directly the dorsal ascending pathways and projecting to the thalamic nuclei, cerebral cortex, and brainstem nuclei, thus stimulating descending motor tracts and interrupting aberrant oscillatory activity in corticobasal nuclei circuits.

The combination of non-invasive neuromodulation with other therapies can enhance the effectiveness of rehabilitation, increasing plasticity and clinical efficacy, offering a greater and more sustained effect than either therapy alone.It's recommended that patients with PD perform a specific exercise for walking, such as treadmill training (tt), that imposes an external rhythm and concentration of attention on gait, acting as an external cue or marker, promoting a more stable gait, reducing gait variability and decreasing risk of falls.

It is proposed, in this study, to develop a new treatment model through the integration of two promising and complementary approaches to improve gait disorders in PD: rTSMS and tt.

Thus, the investigators idealized the realization of the first randomized, double-blind, placebo-controlled, parallel, phase III clinical trial that will evaluate the efficacy of tt associated with rTSMS in patients with PD.

DETAILED DESCRIPTION:
The primary objective is to evaluate the effects of treadmill gait training associated with repetitive transspinal magnetic stimulation on the change in rapid gait speed in Parkinson Disease patients. The investigators hypothesize that the association of repetitive transspinal magnetic stimulation with treadmill gait training should be superior to treadmill gait training alone in improving gait symptoms in patients with PD. Additionally, will be investigated the effects of treadmill gait training associated with repetitive transspinal magnetic stimulation on comfortable gait speed; in clinical and neurophysiological measures; in motor symptoms; in activities of daily living; in the ability to walk (total distance covered); in balance performance; in time to complete the turn; in the severity of the freezing of the gait; in mobility; in the level of physical activity; in the number and fear of falls and in the perception of quality of life of patients with PD. In addition, the possible side effects of the intervention will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18;
* Participants with PD at Hoehn Yahr stages between 2 and 4 (moderate disease) while on-medication (i.e., at the time when their usual dopaminergic medication is clinically effective), whose primary symptom includes gait disturbance (score equal to or greater than 1 in subitem 2.12 of the MSD-UPDRS scale). Patients will be evaluated for the presence of freezing gait (freezing) through the Freezing of Gait Score (FOG-SCORE).
* While on on-medication, be able to walk independently for 30 meters or with a unilateral assistive device.
* Mini Mental State Examination (MMSE) score greater than or equal to 23.
* Sign the informed consent form.

Exclusion Criteria:

* Patients with unstabilized psychiatric comorbidities;
* Individuals who have other neurological disorders, musculoskeletal, orthopedic, cardiovascular and respiratory disorders that may affect the ability to walk on the treadmill will be excluded.
* Individuals with labyrinthine problems, using medication that may interfere with balance and performance in tests and treadmill training will be excluded.
* Individuals who have undergone deep brain stimulation surgery or epidural spinal cord stimulation will be excluded.
* Patients with uncontrolled infection or other uncontrolled pre-existing medical conditions (eg uncontrolled diabetes, high blood pressure, symptomatic lung or heart disease);
* Concomitant treatment with other experimental drugs;
* Pregnant or breastfeeding women.
* Presence of chronic low back and lower limb pain.
* Patients who cannot walk without assistance (cane, crutch, walker) or help from another person.
* Patients with metal implants and a cardiac pacemaker.
* Patient with a history of neurosurgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
10 meter walk test- Fast walking speed | 4 months
  Comparison of the change in fast gait speed between active stimulation and sham stimulation during Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention). Longer time to complete the test results in slower gait speed and worse performance

SECONDARY OUTCOMES:
10 meter walk test- Confortable walking speed | 4 months
  Comparison of the change in confortable gait speed between active stimulation and sham stimulation during Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention). Longer time to complete the test results in slower gait speed and worse performance
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Part II and III | 4 months
  Comparison of change in Unified Parkinson's Disease Rating Scale score part II and III between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention).MDS-PDRS part II is scored from 0 to 52 with higher scores associated with worse motor related daily activities performance. MDS-UPDRS part III is scored from 0 to 132 with higher scores associated with worse motor performance in parkinson related tests.
Freezing of Gait Score- (FOG- SCORE) | 4 months
  Comparison of the change in the severity of gait freezing between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention). The Severity of gait freezing will be evaluated through the Freezing of Gait Score.The score was the sum of the 12 items and it ranges from 0 to 36 points. the higher the score, the worse the performance and severity of gait freezing.
2 Minute Walk Test | 4 months
  Comparison of the change in the Walking capacity (total distance covered) and speed,evaluated through the 2 Minute Walk Test, between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention). A shorter distance covered during 2 minutes results in a slower speed to complete the test and worse performance.
Timed up and Go (TUG) | 4 months
  Comparison of the change in the functional mobility between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention), that will be evaluated through the Timed up and Go test. The time average of two measurements will be calculated. A longer average time to complete the test results in worse performance
Timed up and Go Dual Task (TUG-DT) | 4 months
  Comparison of the change in the Dual-task performance between active stimulation and sham stimulation Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention), that will be evaluated through the Timed up and Go Dual Task test. The time average of two measurements will be calculated. A longer average time to complete the test results in worse performance
Timed 360° turn test | 4 months
  Comparison of the change in the time to complete the turn between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention), that will be evaluated through the Timed 360° turn test. Will be taken 3 measurements for each side and the average of time and of the number of steps required to complete the turn will be calculated. A longer time and a greater number of steps to complete the turn suggests a greater commitment and worse performance
Mini-Balance Evaluation Systems Test (Mini-BESTest) | 4 months
  Comparison of change in the Balance performance between active stimulation and sham stimulation in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention), that will be measured through the Mini-Balance Evaluation Systems Test that includes 14 items scored from 0 to 2, with a maximum score of 28 and a minimum of 0, with a higher score indicating better balance performance.
Freezing of Gait Questionnaire (FOG-Q) | 4 months
  Comparison of change in the subjective perception of the severity and impact of freezing on gait performance between active stimulation and sham stimulation in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention), that will be measured through the Freezing of Gait Questionnaire, that is rated on a 5-point scale (0 to 4), with a total score ranging from 0 to 24. A higher score implies that the individual's gait performance is more affected by freezing
Falls and near falls | 4 months
  The occurrence of falls and near-falls will be investigated through self-report and will be compared between groups in Baseline, right after the end of the 10th session and follow-up (1 month and 3 months post-intervention). The classification of fallers and non-fallers will be obtained.
Human Activity profile (HAP) | 4 months
  Comparison of change in the Level of physical activity between active stimulation and sham stimulation in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention), that will be measured through the Human Activity profile. Tare arranged in ascending order of energy cost.Based on each response, the primary scores are calculated: the maximum activity score (EMA) and the adjusted activity score (EAA).The EAA will be used in this study. The classification of physical activity level will be established through pre-defined cutoff points, with individuals classified as inactive (less than 53), moderately active (between 53 and 74) or active (greater than 74). An increase in the score indicates an improvement in the level of physical activity
Falls Efficacy Scale- International (FES-I) | 4 months
  Comparison of change in the Fear of falls between active stimulation and sham stimulation in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention), that will be measured through the Falls Efficacy Scale- International, that presents questions about the concern with the possibility of falling when performing 16 activities. The total score is calculated by adding the values obtained in each item and can vary from 16 to 64 points, in which the lowest value corresponds to the absence of concern and the highest value to extreme concern regarding falls while carrying out the activities in the questionnaire. Thus, the higher the final score obtained, the lower the self-efficacy related to falls.
Parkinson's Disease Questionnaire -39 (PDQ-39) | 4 months
  The perception of quality of life will be measured in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention) through the Parkinson's Disease Questionnaire -39 which is scored is from 0 to 100, higher values are associated with worse quality of life.
Non-Motor Symptoms Scale (NMSS) | 4 months
  Comparison of change in the Non-Motor Symptoms between active stimulation and sham stimulation in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention) , that will be measured through the Non-Motor Symptoms Scale. The NMSS consists of 30 items and each item's score is based on severity (from 0 to 3) and frequency scores (from 1 to 4).The range for the NMSS total scores is 0-360. Higher scores indicate greater severity of non-motor symptoms
The Parkinson Disease Pain Classification System (PD-PCS) | 4 months
  Comparison of change in pain between active stimulation and sham stimulation in Baseline, 15 days after the end of the 10th session (questionnaire will be applied by phone call at that time) and at follow-up (1 month and 3 months post-intervention), that will be measured through Parkinson Disease Pain Classification System, which scores and classifies parkinson disease-related pain into 3 groups (nociceptive, neuropathic or nociplastic), in relation to intensity, frequency and interference in activities of daily living. Higher scores indicate greater severity of pain
Study of motor evoked potentials (MEPS) | 10 days
  Motor evoked potentials (MEPs) induced by transcranial magnetic stimulation (TMS) will be measured in active and sham stimulation, before the protocol starts and immediately after the 10th session.Thus, in the present study, we sought to evaluate the effects of rTSMS on the characteristics of MEPs at baseline and shortly after the end of the 10th session, evaluating whether rTSMS is a useful technique to facilitate downward impulse and promote motor function in PD.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens G Cury, MD PHD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arii Y, Sawada Y, Kawamura K, Miyake S, Taichi Y, Izumi Y, Kuroda Y, Inui T, Kaji R, Mitsui T. Immediate effect of spinal magnetic stimulation on camptocormia in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2014 Nov;85(11):1221-6. doi: 10.1136/jnnp-2014-307651. Epub 2014 Apr 29. PMID 24780955
- [Background] Chung CL, Mak MK, Hallett M. Transcranial Magnetic Stimulation Promotes Gait Training in Parkinson Disease. Ann Neurol. 2020 Nov;88(5):933-945. doi: 10.1002/ana.25881. Epub 2020 Sep 8. PMID 32827221
- [Background] de Andrade EM, Ghilardi MG, Cury RG, Barbosa ER, Fuentes R, Teixeira MJ, Fonoff ET. Spinal cord stimulation for Parkinson's disease: a systematic review. Neurosurg Rev. 2016 Jan;39(1):27-35; discussion 35. doi: 10.1007/s10143-015-0651-1. Epub 2015 Jul 30. PMID 26219854
- [Background] Fuentes R, Petersson P, Siesser WB, Caron MG, Nicolelis MA. Spinal cord stimulation restores locomotion in animal models of Parkinson's disease. Science. 2009 Mar 20;323(5921):1578-82. doi: 10.1126/science.1164901. PMID 19299613
- [Background] Reis Menezes J, Bernhart Carra R, Aline Nunes G, da Silva Simoes J, Jacobsen Teixeira M, Paiva Duarte K, Ciampi de Andrade D, Barbosa ER, Antonio Marcolin M, Cury RG. Transcutaneous magnetic spinal cord stimulation for freezing of gait in Parkinson's disease. J Clin Neurosci. 2020 Nov;81:306-309. doi: 10.1016/j.jocn.2020.10.001. Epub 2020 Oct 20. PMID 33222935
- [Background] Takakusaki K. Neurophysiology of gait: from the spinal cord to the frontal lobe. Mov Disord. 2013 Sep 15;28(11):1483-91. doi: 10.1002/mds.25669. PMID 24132836
- [Background] Yadav AP, Nicolelis MAL. Electrical stimulation of the dorsal columns of the spinal cord for Parkinson's disease. Mov Disord. 2017 Jun;32(6):820-832. doi: 10.1002/mds.27033. Epub 2017 May 12. PMID 28497877
- [Background] Yang YR, Tseng CY, Chiou SY, Liao KK, Cheng SJ, Lai KL, Wang RY. Combination of rTMS and treadmill training modulates corticomotor inhibition and improves walking in Parkinson disease: a randomized trial. Neurorehabil Neural Repair. 2013 Jan;27(1):79-86. doi: 10.1177/1545968312451915. Epub 2012 Jul 10. PMID 22785003
- [Background] Agari T, Date I. Spinal cord stimulation for the treatment of abnormal posture and gait disorder in patients with Parkinson's disease. Neurol Med Chir (Tokyo). 2012;52(7):470-4. doi: 10.2176/nmc.52.470. PMID 22850494
- [Background] Fenelon G, Goujon C, Gurruchaga JM, Cesaro P, Jarraya B, Palfi S, Lefaucheur JP. Spinal cord stimulation for chronic pain improved motor function in a patient with Parkinson's disease. Parkinsonism Relat Disord. 2012 Feb;18(2):213-4. doi: 10.1016/j.parkreldis.2011.07.015. Epub 2011 Aug 23. No abstract available. PMID 21865071
- [Background] Santana MB, Halje P, Simplicio H, Richter U, Freire MAM, Petersson P, Fuentes R, Nicolelis MAL. Spinal cord stimulation alleviates motor deficits in a primate model of Parkinson disease. Neuron. 2014 Nov 19;84(4):716-722. doi: 10.1016/j.neuron.2014.08.061. Epub 2014 Oct 30. PMID 25447740
- [Background] Pinto de Souza C, Hamani C, Oliveira Souza C, Lopez Contreras WO, Dos Santos Ghilardi MG, Cury RG, Reis Barbosa E, Jacobsen Teixeira M, Talamoni Fonoff E. Spinal cord stimulation improves gait in patients with Parkinson's disease previously treated with deep brain stimulation. Mov Disord. 2017 Feb;32(2):278-282. doi: 10.1002/mds.26850. Epub 2016 Nov 10. PMID 27862267
- [Background] Samotus O, Parrent A, Jog M. Spinal Cord Stimulation Therapy for Gait Dysfunction in Advanced Parkinson's Disease Patients. Mov Disord. 2018 May;33(5):783-792. doi: 10.1002/mds.27299. Epub 2018 Feb 14. PMID 29442369
- [Background] de Lima-Pardini AC, Coelho DB, Souza CP, Souza CO, Ghilardi MGDS, Garcia T, Voos M, Milosevic M, Hamani C, Teixeira LA, Fonoff ET. Effects of spinal cord stimulation on postural control in Parkinson's disease patients with freezing of gait. Elife. 2018 Aug 2;7:e37727. doi: 10.7554/eLife.37727. PMID 30070204
- [Background] Mitsui T, Arii Y, Taniguchi K, Tsutsumi S, Takahara M, Mabuchi M, Sumitomo N, Matsuura M, Kuroda Y. Efficacy of Repetitive Trans-spinal Magnetic Stimulation for Patients with Parkinson's Disease: a Randomised Controlled Trial. Neurotherapeutics. 2022 Jul;19(4):1273-1282. doi: 10.1007/s13311-022-01213-y. Epub 2022 Jun 27. PMID 35759108